CLINICAL TRIAL: NCT05267314
Title: Impact of External Pharyngeal Exerciser on Dysphagia in Patients With Pharyngeal Weakness
Brief Title: External Pharyngeal Exerciser for Dysphagia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Anisa Shaker, Associate Professor of Medicine, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-16-00374
Record Dates: First submitted 2022-01-24; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Pharyngeal Dysphagia; Dysphagia; Oral Pharyngeal Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard therapy (No Intervention): standard therapy
- exerciser and standard therapy (Experimental): exerciser and standard therapy
  Interventions: Device: pharyngeal exerciser + standard therapy

INTERVENTIONS:
Device: pharyngeal exerciser + standard therapy — Use of Pharyngeal exerciser
  Arms: exerciser and standard therapy

SUMMARY:
Pharyngeal muscle weakness and dysphagia is common in individuals post-stroke or with Parkinson's disease and in individuals with head/neck cancer who have undergone surgery and/or radiation therapy. Therapeutic options for these patients are limited. This pilot study is intended to assess the feasibility, safety, and efficacy of the External Pharyngeal Exerciser (EPE) on patients with pharyngeal dysphagia receiving swallow therapy. Feasibility will be assessed by patient acceptance and practice records. Safety will be compared between groups to test whether there is an increased risk of the EPE versus standard therapy.

DETAILED DESCRIPTION:
Pharyngeal dysphagia is incredibly common in individuals who suffer from neurological disorders such as stroke or Parkinson's disease and in individuals with head/neck cancer who have undergone surgery and/or radiation therapy. The pharyngeal muscles in these patients are weak. Other than standard patient-driven swallow therapy, the therapeutic options for these patients are limited. Response to standard patient-drive therapy is variable and dependent on a variety of factors including the muscles most affected by the underlying disorder and patient motivation. This pilot study is intended to assess the feasibility, safety, and efficacy of the External Pharyngeal Exerciser (EPE) on patients with pharyngeal dysphagia receiving swallow therapy. Feasibility will be assessed by patient acceptance and practice records. Safety will be compared between groups to test whether there is an increased risk of the EPE versus standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pharyngeal dysphagia diagnosed with validated questionnaire and modified barium swallow. Participants must be at least 18 years of age or older.
* Pharyngeal dysphagia secondary to central neurological disorder such as Parkinson's disease or stroke
* Pharyngeal dysphagia head/neck cancer secondary to surgery/radiation
* Pharyngeal dysphagia secondary to elderly age > 65

Exclusion Criteria:

* Carotid artery bruit or carotid vascular disorders
* Muscle diseases like muscular dystrophies, myopathies
* Neuro-muscular junction disorders myasthenia gravis, Eaton-Lambert disorders
* Current esophageal symptoms like heartburn, dysphagia, chest pain or regurgitation
* Autonomic dysfunction
* Pregnancy or lactation
* Advanced uncontrolled medical disorders (COPD, congestive heart failure, cirrhosis, cancer, chronic renal failure, etc)
* Medically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-12-06 (Estimated); Study Completion 2022-12-06 (Estimated)

PRIMARY OUTCOMES:
Determine the number of adverse events associated with EPE | 1 year
  The aim is to determine whether there are any risks associated with the use of the EPE. There are no known risks to placing external pressure to the larynx. However, there is the possibility that the participant may experience discomfort such as rash or may not be able to tolerate the minimal pressure associated with the exerciser. The participant will be evaluated every two weeks by the study physician and reports of adverse events will be recorded. If the participant experiences difficulty in tolerating the minimal pressure, the study will be stopped.
Determine efficacy as assessed by validated pharyngeal dysphagia questionnaire EAT-10 | 1 year
  Subjective evaluation of participant response to an External Pharyngeal Exerciser with a validated pharyngeal dysphagia questionnaire (EAT-10) administered as standard of care before and after therapy (scores 1-10, with higher scores mean worse outcome).
Determine efficacy: effect of EPE on swallowing via effects on pyriform sinus and vallecular residue height and width | 1 year
  To objectively define pharyngeal response to External Pharyngeal Exerciser with Modified Barium swallow before and after therapy: To determine if application of pharyngeal exerciser changes swallowing as evidenced by reduction in height and width of pyriform sinus and vallecular residue using fluoroscopy study.
Determine efficacy: effect of EPE on swallowing via effects on routinely measured markers of deglutition (penetration-aspiration scale, larynx and hyoid anterior/superior excursion; UES diameter, and pharyngeal transit time) | 1 year
  To objectively define pharyngeal response to External Pharyngeal Exerciser with Modified Barium swallow before and after therapy: To determine if application of pharyngeal exerciser changes deglutition as noticed by 1) change in aspiration and penetration measured by Rosenbek's penetration-aspiration scale; 2) change in anterior and superior excursion of larynx and hyoid; 3) change in AP and Lateral diameter of UES; 4) change in pharyngeal transit time.

SECONDARY OUTCOMES:
Physiologic change in swallow performance identified on routine Modified barium swallow | 1 year
  Physiologic changes in swallow performance: oral-motor strength, vocal cord adduction with various food consistencies, presence of penetration/aspiration, length of anterior and superior excursion of larynx, pharyngeal transit time, presence and width of vallecular/piriform residue. Poor anterior or superior excursion of larynx, diminished AP and lateral diameter of UES, presence of residue, penetration/aspiration suggests pharyngeal dysphagia. These measurements will be combined/aggregated to arrive at one reported value.

CONTACTS AND LOCATIONS:
Locations (1):
- Anisa Shaker, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No